CLINICAL TRIAL: NCT00844064
Title: An Open-Label, Multicenter Dose-Escalation Study to Evaluate the Safety and Tolerability of AP 12009 (Trabedersen), Administered Intravenously in Patients With Advanced Tumors Known to Overproduce TGF-β2.
Brief Title: Safety and Tolerability of AP 12009, Administered I.V. in Patients With Advanced Tumors Known to Overproduce TGF-beta-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isarna Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP 12009-P001
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Neoplasms; Melanoma; Colorectal Neoplasms
Keywords: Pancreatic cancer; Metastatic melanoma; Advanced tumor; Targeted therapy; Antisense; Transforming Growth Factor beta 2; Dose escalation
MeSH Terms: conditions — Pancreatic Neoplasms; Melanoma; Colorectal Neoplasms | interventions — Trabedersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AP 12009 (Experimental)
  Interventions: Drug: AP 12009

INTERVENTIONS:
Drug: AP 12009 — Initial scheme: AP 12009 (trabedersen), dose escalation scheme, continuous intravenous infusion (7 days), every other week, up to 10 cycles.
  Modified scheme: AP 12009 (trabedersen), dose escalation scheme, continuous intravenous infusion (4 days), every other week, up to 10 cycles

SUMMARY:
In this national Phase I dose-escalation study the safety and tolerability of AP 12009 is evaluated in adult patients with advanced tumors known to overproduce TGF-β2, who are not or no longer amenable to established therapies.

DETAILED DESCRIPTION:
The purpose of this dose-finding study is to evaluate the safety and tolerability of AP 12009. Two fixed dose-escalation schemes with predefined steps and increasing increments have been selected to determine the maximum tolerated dose (MTD) as well as the dose-limiting toxicity (DLT). At least two cycles of AP 12009 are administered intravenously in adult patients with no further acknowledged treatment options.

AP 12009 (trabedersen) is a phosphorothioate antisense oligodeoxynucleotide specific for the mRNA of human Transforming Growth Factor beta 2 (TGF-beta-2). The growth factor TGF-beta plays a key role in malignant progression of various tumors by inducing proliferation, invasion, metastasis, angiogenesis, and escape from immunosurveillance. In patients with pancreatic cancer, colorectal cancer, and metastatic melanoma the TGF-beta-2 overexpression is associated with disease stage, clinical prognosis, and the immunodeficient state of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age: 18-75 years.
3. Male or non-pregnant, non-lactating female.
4. a.Pancreatic cancer: Histologically or cytologically confirmed diagnosis, stage IVA or IVB (AJCC, 1997).

   b. Melanoma: Histologically or cytologically confirmed diagnosis, stage III or IV (AJCC, UICC).

   c. Colorectal cancer: Histologically or cytologically confirmed diagnosis, stage III or IV (AJCC, UICC), excluded from the last cohort.
5. Patient is not or no longer amenable to established forms of therapy.
6. At least one measurable lesion.
7. Karnofsky performance status of at least 80%.
8. Recovery from acute toxicity caused by any previous therapy.
9. Adequate organ function as assessed by the following laboratory values:

   * Serum creatinine and urea < 2 times the upper limit of normal (ULN).
   * ALT and AST < 3 ULN (in case of a liver metastasis: < 5x ULN); alkaline phosphatase < 3 ULN; and bilirubin < 2.5 mg/dL.
   * Prothrombin time < 1.5 INR and PTT < 1.5 times the upper limit of normal.
   * Hemoglobin > 9 g/dL.
   * Platelets > 100 x 10E9/L.
   * WBC > 3.0 x 10E9/L.
   * Absolute Neutrophil Count (ANC) > 1.5 x 10E9/L.

Exclusion Criteria:

1. Patient unable to comply with the protocol regulations.
2. Pregnant or lactating female.
3. Antitumor radiation therapy within 12 weeks, tumor surgery within 4 weeks or any other therapy with established antitumor effects within 2 weeks prior to study entry.
4. The patient takes or is likely to need other prohibited concomitant medication. Administration of corticosteroids should be strictly avoided during the course of the study.
5. Patient's participation in another clinical trial with investigational medication within 30 days prior to study entry.
6. History of brain metastases. In the case of suspected brain metastases a CT scan of the skull will be performed (not mandatory in asymptomatic patients).
7. Clinically significant cardiovascular abnormalities such as refractory hypertension, congestive heart failure, unstable angina, or poorly controlled arrhythmia, or a myocardial infarction within 6 months prior to treatment.
8. Gastric or duodenal ulcers within 6 months before study entry or is at risk of gastrointestinal ulceration due to high consumption of NSAIDs.
9. An active infection with HIV, HBV, or HCV.
10. Clinically significant acute viral, bacterial, or fungal infection.
11. Acute medical problems that may be considered to become an unacceptable risk, or any conditions that might be contraindications for starting study treatment.
12. History of allergies to reagents used in this study.
13. Drug abuse or extensive use of alcohol.
14. Significant psychiatric disorders/ legal incapacity or limited legal capacity.
15. History of Long QT Syndrome or QTc time ≥ 480 msec in screening/baseline ECGs. The average QTc time is to be calculated from three separate ECGs performed prior to start of infusion: two ECGs performed at Screening/Baseline (with a minimum 1-hour interval in between) and one performed within 1 hour prior to start of infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) as well as the dose-limiting toxicity (DLT) of two cycles of AP 12009 administered intravenously at weekly intervals and for four days every other week.

SECONDARY OUTCOMES:
To determine the safety and tolerability of AP 12009 administered intravenously at weekly intervals and for four days every other week.
To assess the plasma pharmacokinetic profile of AP 12009 administered intravenously at weekly intervals and for four days every other week.
To establish a suitable determination method and to assess the urine pharmacokinetic profile of AP 12009 administered intravenously for four days every other week.
To determine the effect of AP 12009 administered intravenously at weekly intervals and for four days every other week on TGF-β2 plasma concentration levels.
To determine the potential antitumor activity of AP 12009 administered intravenously at weekly intervals and for four days every other week, as assessed by the effect on tumor size and tumor markers.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Oettle, MD, Study Chair — Charité Berlin Campus Virchow-Klinikum
Locations (10):
- Germany (10):
  - Universitätsmedizin Berlin Charité, Berlin
  - Universitätsklinik und Poliklinik für Innere Medizin I, Halle
  - Hautklinik der Ruprecht-Karls-Universität Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Krankenhaus rechts der Isar, II. Medizinische Klinik und Poliklinik, München
  - Universität Münster, Klinik und Poliklinik für Hautkrankheiten, Münster
  - Klinik und Poliklinik für Innere Medizin I, Regensburg
  - Klinik und Poliklinik für Dermatologie, Regensburg
  - Universitäts-Hautklinik, Sektion Dermatologische Onkologie, Tübingen
  - Universitätsklinikum Ulm, Zentrum für Innere Medizin, Ulm